CLINICAL TRIAL: NCT05313724
Title: Mind-body Online Therapy in a Somatic Setting - a Randomized-controlled, Two-arm, Monocentric Study in Gynecological Oncology
Brief Title: Mind-body Online Therapy in Gynecological Oncology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Katja Haemmerli Keller (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor-Investigator, Katja Haemmerli Keller, Principal Investigator, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022-00174
Record Dates: First submitted 2022-03-11; First posted 2022-04-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Gynecologic Cancer
Keywords: Mind; Body; MBM; Mind Body Medicin; Online Therapy; Online-Therapie; Internettherapie; Internet Therapy; Selbsthilfeintervention; Onkologie; Oncology; Krebs; Cancer; Gynäkologie; Gynecology; Frauenklinik; Frauenheilkunde; Psychosomatik; Psychosomatics; Psychotherapie; Psychotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind-Body Online Therapy (Experimental)
  Interventions: Other: Mind-Body Online Therapy
- TAU (treatment as usual) (No Intervention)

INTERVENTIONS:
Other: Mind-Body Online Therapy — There are 8 different modules (e.g. relaxation, mindfulness, stress management, disease management, nutrition and exercise behavior) with a mind-body focus available for the patients to independently (time, location) work on.
  Arms: Mind-Body Online Therapy

SUMMARY:
In this randomized-controlled two-arm monocentric study with three measurement time points, the effectiveness and feasibility of an internet-based, therapist-guided mind-body self-help intervention for gynecological cancer patients with primary diagnoses is examined. Different modules (e.g., relaxation, mindfulness, stress management, disease management, nutrition and exercise behaviors) with a mind-body focus are available for the patients. The goal of the intervention is to improve or maintain the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Oncologic disease: first diagnosed; within the first 12 weeks of diagnosis, first-line treatment (either systemic treatment - including chemotherapy, hormonal therapy or targeted therapy - or radiotherapy), Notes: (1) Patients treated for first recurrence of a tumor previously treated with curative intent are also eligible. (2) Psychological distress is taken into account by stratification according to the stress thermometer. In research, this procedure corresponds to the current state-of-the-art. Individual subgroups (e.g. cancer stages) can then be studied post-hoc.
* Sufficient computer skills and internet access
* Availability of an emergency address
* Written informed consent by signing the informed consent form

Exclusion Criteria:

* Patient unable to provide written informed consent by signing informed consent form
* Insufficient knowledge of German
* Moderate to severe depressive symptomatology (BDI > 18; HAM-D17 ≥ 17) during T1 survey
* Suicidality (BDI suicidality item > 1; HAM-D17 suicidality item ≥ 2) in the context of the T1 survey
* Diagnosis of psychotic, bipolar, or other serious mental or somatic disorder requiring immediate treatment
* Male breast cancer patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety and depression | Changes between week 0, 8, 16
  German version of the questionnaire "Hospital Anxiety and Depression Scale" (HADS; (Herrmann et al., 1995; Herrmann-Lingen et al., 2011)
Depression (external assessment) | Changes between week 0, 8, 16
  German version of the questionnaire "Hamilton Depression Scale" (HAM-D17; Hamilton, 1960; Hamilton, 1986)
Somatization | Changes between week 0, 8, 16
  German version of the questionnaire "Patient Health Questionnaire" (PHQ-9; Gräfe et al., 2004; Kroenke et al., 2010)
General distress | Week 0, Week 8, Week 16
  German version of the questionnaire "Distress Thermometer" (BTH; Mehnert et al., 2006)
Psychological stress | Changes between week 0, 8, 16
  German version of the questionnaire "Symptom Checklist" (SCL-K11; Franke, 2001; Franke, 2002)
Impairment from cancer therapy | Changes between week 0, 8, 16
  German version of the questionnaire "Functional Assessment of Cancer Therapy" (FACT-G; Cella & Bonomi, 1996; Cella et al., 1993)
Insomnia (Severity) | Changes between week 0, 8, 16
  German version of the questionnaire "Insomnia Severity Index" (ISI; Morin, 1993)
Sleep quality | Changes between week 0, 8, 16
  German version of the questionnaire "Pittsburgh Sleep Quality Index" (PSQI; Buysse et al., 1989; Carpenter & Andrykowski, 1998)
Health-related quality of life | Changes between week 0, 8, 16
  German version of the questionnaire "Short Form 12" (SF-12; Morfeld et al., 2012)
SpO2 [%] | Changes between week 0, 8, 16
  Sleep diagnostic system "WatchPAT" (Neumedpro, Neuwirth Medical Products, 2021)
Peripheral arterial tone (PAT) [mmHG] | Changes between week 0, 8, 16
  Sleep diagnostic system "WatchPAT" (Neumedpro, Neuwirth Medical Products, 2021)

SECONDARY OUTCOMES:
Feasibility of the intervention (Patient-therapist relationship) | Changes between week 8, 16
  German version of the questionnaire "Working Alliance Inventory - Short Revised" (WAI-SR; Wilmers et al., 2008)
Feasibility of the intervention (Usability) | Changes between week 8, 16
  German version of the questionnaire "System Usability Scale" (SUS; Brooke, 1996)
Feasibility of the intervention (Patient satisfaction) | Changes between week 8, 16
  German questionnaire "Patient Satisfaction" (ZUF-8; Schmidt & Wittmann, 2002)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Psychosomatic Medicine and Consultation-Liaison Psychiatry, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No